CLINICAL TRIAL: NCT05791591
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Study to Evaluate Safety and Efficacy of Orally Administered NUV001 Nutraceutical Supplement in Sickle Cell Disease Patients.
Brief Title: Safety and Efficacy of Orally Administered NUV001 Nutraceutical Supplement in Sickle Cell Disease Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LGD (Industry)
Collaborators: ProRelix Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LGD-NUV001-CT01-22; LGD-CLI-006 (Other: LGD)
Record Dates: First submitted 2023-02-21; First posted 2023-03-30 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Sickle Cell Disease
Keywords: Hb-SS; Hb S/β0-Thal
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NUV001 - IR (Experimental): Sickle cell disease patients receiving NUV001 Immediate release gel capsule formulation
  Interventions: Dietary Supplement: NUV001 - IR
- NUV001 - GR (Experimental): Sickle cell disease patients receiving NUV001 Gastro resistant gel capsule formulation
  Interventions: Dietary Supplement: NUV001 - GR
- Placebo (Placebo Comparator): Sickle cell disease patients receiving Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NUV001 - IR — Daily supplementation with 1000 mg of NUV001 (in two administration orally) immediate release gel capsule formulation for 90 days in total
  Arms: NUV001 - IR
Dietary Supplement: NUV001 - GR — Daily supplementation with 1000 mg of NUV001 (in two administration orally) gastro resistant gel capsule formulation for 90 days in total
  Arms: NUV001 - GR
Dietary Supplement: Placebo — Placebo containing starch Powder (1000 mg, daily in two administration orally for 90 days)
  Arms: Placebo

SUMMARY:
A total of 170 patients male or female who are carrying SS or Sbeta0 versions of the beta globin gene will be included in the study. The subjects will be assigned with 1:1:1 ratio of either NUV001 Immediate release IR or NUV001 Gastro resistant GR or Placebo. The treatment duration of the study will be 90 days which has in total 5 visits. The primary end point of this study is to check the safety and tolerance of the orally administered nutraceutical supplement. This endpoint will be checked by assessing the Adverse events, Vital signs of the subject and the Change in hematological parameters from Baseline to Final visit.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women over 18 to 65 years, both inclusive.
2. Non-smokers.
3. BMI > 18 kg/m2
4. Patients diagnosed with sickle cell disease (documented by haemoglobin electrophoresis) and carrying SS or Sbeta0 versions of the beta globin gene (documented by genotyping, known through medical history).
5. Haemoglobin levels between 5.5 and 10.5 g/dl during Screening (for newly diagnosed or patients not on any treatment for SCD).
6. If the patient has been treated with an anti-sickling agent within three months of the Screening visit, the therapy must have been continuous for at least three months with the intent to continue for the duration of the study.
7. Available to attend on an outpatient basis for visits provided for in the protocol and able to complete the data collection documents (compliance and quality of life scale)
8. Patient or the patient's legally authorized representative has given written informed consent.

Exclusion Criteria:

1. Patients with known or suspected allergy to any ingredient of the food supplement
2. Patient having consumed vitamin or food supplements containing NAD+ precursors (niacin, tryptophan, nicotinamide, NMN, NR etc...) during the month before selection.
3. Patient has a significant medical condition that required hospitalization (other than sickle cell crisis) within two months of the screening visit.
4. Patient has prothrombin time INR > 2.0.
5. Patient has serum albumin less than 3.0 g/dl.
6. Patient has received any blood products within three months of the Screening visit.
7. Patients hospitalized for acute vaso-occlusive crisis within one month of the Screening visit.
8. Patient has clinically significant, cardiovascular or liver disease or renal insufficiency or lymphopenia , evident in medical history (with clinically significant abnormal results on the Screening bioassays for eg.: Complete blood count, Aspartate transaminases, Alanine transaminases, Gamma glutamyl transferase, Alkaline Phosphatase, Bilirubin, Creatinine, Creatinine Phosphokinase, Blood Glucose, HbA1c, Lipid Profile).
9. Patient with diagnosed cancer in the past 2 years.
10. Patients participating simultaneously in another clinical research protocol or having recently participated in another research for which the exclusion period has not been completed.
11. Pregnant, lactating or parturient women.
12. Persons deprived of their liberty by a judicial or administrative decision, hospitalized without consent or admitted to a health or social establishment for purposes other than that of research.
13. Majors under legal protection or unable to express their consent.
14. People in an emergency situation unable to express their prior consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by subject incident of treatment-emergent adverse events | between Day 0 and Day 30
  Subject incidence of treatment-emergent adverse events
Safety as measured by subject incident of treatment-emergent adverse events | between Day 0 and Day 60
  Subject incidence of treatment-emergent adverse events
Safety as measured by subject incident of treatment-emergent adverse events | between Day 0 and Day 90
  Subject incidence of treatment-emergent adverse events
Safety as measured by subject incident of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete Blood Count (absolute counts and %), Random blood glucose concentration and Serum concentrations in Calcium, Electrolytes, Protein, Albumin, Alkaline Phosphatase, Bilirubin, Blood urea nitrogen, Creatinine, Aspartate Aminotransferase, Alanine Aminotransferase)
Safety as measured by subject incident of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 60
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete Blood Count (absolute counts and %), Random blood glucose concentration and Serum concentrations in Calcium, Electrolytes, Protein, Albumin, Alkaline Phosphatase, Bilirubin, Blood urea nitrogen, Creatinine, Aspartate Aminotransferase, Alanine Aminotransferase)
Safety as measured by subject incident of treatment-emergent clinically significant changes in clinical laboratory safety tests | between Day 0 and Day 90
  Subject incidence of treatment-emergent clinically significant changes in clinical laboratory safety tests (Complete Blood Count (absolute counts and %), Random blood glucose concentration and Serum concentrations in Calcium, Electrolytes, Protein, Albumin, Alkaline Phosphatase, Bilirubin, Blood urea nitrogen, Creatinine, Aspartate Aminotransferase, Alanine Aminotransferase)
Safety as measured by subject incident of treatment-emergent clinically significant changes in vital signs | between Day 0 and Day 30
  Subject incidence of treatment-emergent clinically significant changes in vital signs (Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg), Pulse Rate in beats per minute (bpm), Respiration Rate in number of breaths per minute and Body temperature in Celsius)
Safety as measured by subject incident of treatment-emergent clinically significant changes in vital signs | between Day 0 and Day 60
  Subject incidence of treatment-emergent clinically significant changes in vital signs (Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg), Pulse Rate in beats per minute (bpm), Respiration Rate in number of breaths per minute and Body temperature in Celsius)
Safety as measured by subject incident of treatment-emergent clinically significant changes in vital signs | between Day 0 and Day 90
  Subject incidence of treatment-emergent clinically significant changes in vital signs (Systolic and Diastolic Blood Pressure in millimeters of mercury (mmHg), Pulse Rate in beats per minute (bpm), Respiration Rate in number of breaths per minute and Body temperature in Celsius)

SECONDARY OUTCOMES:
Change in the % of F-hemoglobin positive cells | Day 0, Day 30, Day 60, Day 90
Change in F-Hb content in RBCs | Day 0, Day 30, Day 60, Day 90
  % of total hemoglobin measured by HP-LC
Change in RBC sickling | Day 0, Day 30, Day 60, Day 90
  % of circulating irreversibly sickled cells
Change in hematocrit | Day 0, Day 30, Day 60, Day 90
  % of RBC in blood
Change in indirect bilirubin level | Day 0, Day 30, Day 60, Day 90
  Indirect bilirubin level expressed in mg/dL
Change in reticulocyte level | Day 0, Day 30, Day 60, Day 90
  reticulocytes count expressed in percentage of red blood cells
Change in serum lactate dehydrogenase level | Day 0, Day 30, Day 60, Day 90
  Serum lactate dehydrogenase expressed in international units per liter (IU/L)
ASCQ-Me Questionnaire (Adult Sickle Cell Quality of Life Measurement Information System) | Day 0, Day 30, Day 60, Day 90
  Questionnaire on acute and/or chronic pain, energy level, usage of pain medications and activity levels
Change in pain perception | Day 0, Day 30, Day 60, Day 90
  Evaluation of pain intensity for each body location (using a numeric pain rating scale from 0, no pain to 10 worst possible pain)
Pain relief assessment | Day 0, Day 30, Day 60, Day 90
  Evaluation and evaluation of pain relief (pain relief scale in percent from 0%, no relief to 100% complete relief)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Canault, PhD, Study Director — LGD
Locations (8):
- India (8):
  - Aman Hospital and Research Center, Vadodara, Gujarat
  - Kingsway Hospital, Nagpur, Maharashtra
  - Sai Krupa Hospital & Research Centre, Ahmedabad
  - Thalassemia & Sickle Cell Society, Hyderabad
  - Index Medical College, Indore
  - NRSMC Hospital, Kolkata
  - Arihant Hospital, Nagpur
  - Shalinitai Meghe Hospital & Research Centre, Nagpur

IPD SHARING:
Plan to Share IPD: No